CLINICAL TRIAL: NCT05664867
Title: Developing and Optimizing Best Practice Solutions for Implementation of Population Based Cancer Genetic Services in Federally Qualified Health Centers
Brief Title: Implementation of Population Cancer Genetic Services in Federally Qualified Health Centers (FQHC)
Acronym: TestMiGenes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Pamela Ganschow, Principal Investigator, University of Illinois at Chicago
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 2022-1151
Record Dates: First submitted 2022-10-31; First posted 2022-12-27 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-10

CONDITIONS: Hereditary Cancer Syndrome
MeSH Terms: conditions — Neoplastic Syndromes, Hereditary

STUDY DESIGN:
Intervention Model Description: clinical trial with a hybrid effectiveness-implementation quasi-experimental design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MGT (Mainstream Genetic Testing) Model (Experimental): The mainstream genetic testing (MGT) model of cancer genetic services involves a non-genetics healthcare provider, such as the primary care provider, who engages patients in the counseling, consenting, and ordering of genetic testing. The provider/care team discloses the genetic test results and refers patients for genetic counseling only when genetic test results are abnormal. By eliminating the pre- and post-test counseling visits with a genetics provider, the MGT model has the potential to provide scalable access to genetic services.
  Interventions: Other: Mainstream Genetic Testing Model
- SOC (Standard of Care) Model (Active Comparator): The enhanced standard of care model (SOC+) is the current referral model of cancer genetic services delivery with an enhancement to include screening for and resources to address health literacy. This model begins with a health care provider's recognition, identification and then referral of a patient to a genetic counselor where genetic testing takes place if appropriate. This model is time- and resource- intensive and may not be scalable.
  Interventions: Other: Enhanced Standard of Care Model

INTERVENTIONS:
Other: Mainstream Genetic Testing Model — Mainstream Genetic Testing Model of Cancer Genetics Service Delivery
  Other Names: MGT
  Arms: MGT (Mainstream Genetic Testing) Model
Other: Enhanced Standard of Care Model — Enhanced Standard of Care Model of Cancer Genetic Service Delivery
  Other Names: SOC+
  Arms: SOC (Standard of Care) Model

SUMMARY:
The goal of this clinical trial is for researchers to compare the effectiveness of a mainstreamed model of genetic testing (MGT) with an enhanced standard of care model (SOC+) on the uptake of genetic testing among at-risk patients in an urban Federally Qualified Health Center (primary care) setting using a hybrid-effectiveness study design.

Aim 1 is to compare the effectiveness of MGT and SOC+ interventions on the uptake of genetic testing among patients receiving primary care in an urban federally qualified health center (FQHC) system using a randomized trial study design. The hypothesis is that the uptake of testing will be higher among patients receiving services through the MGT compared with the SOC+ model.

Aim 2 is to evaluate the implementation outcomes (acceptability, feasibility and sustainability) and the barriers and facilitators of cancer genetic service delivery approaches within primary care at FQHCs via qualitative interviews with patients, primary care providers and clinic staff, and organizational leaders, guided by the Explore, Prepare, Implement, Sustain (EPIS) implementation framework.

The study will take place at four community health clinics that are part of a Federally Qualified Health Center (FQHC) network in Chicago. Each clinic will use one of two ways of providing cancer genetic services: an enhanced standard of care model that includes patient navigation support (SOC+), or a mainstream genetic testing model (MGT) in which primary care providers offer testing directly. Information such as patients' demographic characteristics, referrals for genetic counseling, completion of genetic testing, and how long it takes to complete testing will be collected from clinic records. Patients, healthcare providers, and clinic staff will also be invited to take part in interviews to share their experiences and perspectives on how each model worked in practice.

DETAILED DESCRIPTION:
More than 15 years after the release of evidence-based guidelines recommending hereditary cancer risk assessment and testing for at-risk individuals, fewer than one in five eligible patients receive this care. Utilization of cancer genetic services remains substantially lower among racial and ethnic minority populations. Addressing inequities in access to these services is essential, as approximately 10 to 15 percent of cancers are linked to inherited mutations, and early identification of high-risk individuals can support prevention and early detection strategies that reduce disparities in cancer outcomes.

Multiple social determinants of health (SDoH) contribute to limited access to genetic services among underserved populations. At the clinic level, many community health centers have limited capacity to systematically identify at-risk patients, employ few or no genetic specialists, and must rely on external systems for genetic counseling and testing. At the provider level, primary care clinicians often report low confidence and limited training in cancer genetics, while genetic specialists may have limited presence or integration in these care settings. At the patient level, structural, economic, and cultural barriers continue to restrict engagement in genetic testing and counseling.

This project will evaluate and compare two models of cancer genetic service delivery in primary care to improve equitable access among patients served by Federally Qualified Health Centers (FQHCs). The enhanced standard of care model (SOC+) uses universal electronic hereditary cancer risk assessment (HCRA) to identify eligible patients, combined with patient navigation to address individual barriers such as financial concerns and literacy needs. The mainstream genetic testing model (MGT) embeds genetic testing directly into primary care visits, allowing patients to receive education, counseling, and test ordering from their primary care provider without referral to specialty care.

Aim 1: Compare the effectiveness of MGT and SOC+ on uptake of genetic testing among minority patients receiving primary care within an urban FQHC system.

Aim 2: Evaluate implementation outcomes (acceptability, feasibility, and sustainability) and identify barriers and facilitators to cancer genetic service delivery in primary care using qualitative interviews with patients, providers, and clinic staff, guided by the Exploration, Preparation, Implementation, Sustainment (EPIS) framework.

A quasi-experimental design will be used across four FQHC clinics, with each clinic assigned to one of the two models, two SOC+ and two MGT. Demographic and service utilization data, including referrals, testing completion, and time-to-test intervals, will be collected from the electronic medical record. Semi-structured interviews with patients, providers, and staff will further explore experiences and perceptions of each model.

This work will generate actionable evidence on scalable and sustainable approaches to delivering guideline-based genetic services in underserved primary care settings. Findings will inform best practices to reduce inequities in access to precision cancer prevention and early detection services.

ELIGIBILITY:
Aim 1 and 2 Inclusion Criteria for patients

1. Adults age 25+
2. English speaking
3. Identified as eligible for cancer genetic testing for a hereditary breast or colon cancer syndrome (e.g., BRCA, Lynch or familial polyposis syndrome) as defined by NCCN criteria45-46
4. Screened positive and agreed to have study staff contact them in the future to participate in virtual/telephone interviews about their experiences with cancer genetics services.
5. Patient receiving care from one of the 4 Federally Qualified Health Center clinics enrolled in the clinical trial

Exclusion Criteria:

1. Did not meet the inclusion criteria
2. Did not screen positive on HCRA and/ or did not agree to have study staff contact them in the future to participate in virtual/telephone interviews about their experiences with cancer genetics services.
3. Not a patient receiving care from the one of the clinics enrolled in the clincial trial

Aim 2

Inclusion Criteria for Providers/Staff:

1. Provider or staff member at one of the 4 clinics participating in the clinical trial
2. English speaking

Exclusion Criteria:

1. Does not meet inclusion criteria above

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Uptake of genetic testing | 2 years
  compare the uptake of genetic testing among patients in both models of cancer genetic delivery who screen positive on hereditary cancer risk asserssment (HCRA)

SECONDARY OUTCOMES:
Time to genetic testing | 2 years
  Time from screening positive on HCRA to genetic testing
Evaluate the implementation outcomes (acceptability, feasibility and sustainability) and the barriers and facilitators of cancer genetic service delivery approaches within primary care at FQHCs | 2 years
  Qualitative interviews with patients and providers in the clinical trial, guided by the Explore, Prepare, Implement, Sustain (EPIS) implementation framework.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Illinois Cancer Center, Chicago, Illinois, United States